CLINICAL TRIAL: NCT02721316
Title: Randomized Study of Ambulatory Monitoring Nurse Under the Prevention of Recurrent Suicidal
Brief Title: Outpatient Nurse Monitoring Under the Prevention of Recurrent Suicidal
Acronym: SIPRéS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UF9533
Record Dates: First submitted 2016-03-08; First posted 2016-03-29 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2022-02

CONDITIONS: Mood Disorder; Reactive Depression
MeSH Terms: conditions — Mood Disorders; Adjustment Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supported with intensive nursing follow (Experimental): Supported with intensive nursing follow post hospitalization the team of hospital output of the unit to 12 weeks after discharge. These interviews will be conducted at the hospital, at home or by phone and their pace will be adjusted according to the patient's condition. The expected duration of close outpatient follow-up is of maximum 3 months.
  Interventions: Other: Supported with intensive nursing follow post hospitalization
- usual care (No Intervention): For control patients, monitoring will be identical to their usual care as part of their pathology.

INTERVENTIONS:
Other: Supported with intensive nursing follow post hospitalization — Intensive nursing follow post - hospitalization
  Arms: Supported with intensive nursing follow

SUMMARY:
To evaluate the impact of a specific nursing management (personalized and close, through consultation at the hospital, at home or by phone) monitoring in post-hospitalization, the suicide attempt of recurrence and suicidal crisis, in the year following a suicide attempt in patients suffering from a mood disorder (unipolar or bipolar) or reactive depression.

DETAILED DESCRIPTION:
Main objective: To evaluate the impact of a specific nursing management (personalized and close, through consultation at the hospital, at home or by phone) monitoring in post-hospitalization, the suicide attempt of recurrence and suicidal crisis, in the year following a suicide attempt in patients suffering from a mood disorder (unipolar or bipolar) or reactive depression.

Secondary objectives:

Studying during the year following the suicide attempt index, the impact of this device on:

* The frequency and intensity of suicidal ideation
* the spontaneous use of emergency care
* the death rate from suicide and other causes
* the cumulative duration of hospitalization for suicidal behavior
* The patient's quality of life
* the number of patients lost to at the end of search

Studying patient compliance with intensive nursing monitoring program.

To study the role of the nurse to determine the factors that promote the construction of a therapeutic alliance.

Establish a mapping of needs and resources suicidal patient for nursing care in post-emergency.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a mood disorder (unipolar or bipolar) or reactive depression whose reason for hospitalization in the Psychiatric Emergency Unit Post has attempted suicide

Exclusion Criteria:

* Patients with bipolar disorder, current episode manic in
* Patient Hospitalized full-time (for high suicide risk incompatible with an output of emergencies or clinical transfer) within 3-5 days of the TS
* Patient suffering from a somatic pathology associated with the prognosis is committed in the short term.
* Patients suffering from a neurodegenerative pathology of dementia or pre-dementia types.
* Homeless Patient

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Change the suicidal rate of recurrence between patients with intensive nursing follow post - hospitalization and patients with usual care | Day 3rd, 6rd day, 3 weeks, 6 weeks and 12 week after emergency exit

SECONDARY OUTCOMES:
Change in the number of emergency hospitalization for suicidal crisis without acting out between patients with intensive nursing follow post - hospitalization and patients with usual care | Day 3rd, 6rd day, 3 weeks, 6 weeks and 12 week after emergency exit

CONTACTS AND LOCATIONS:
Overall Officials: Grégory Mykolow, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided